CLINICAL TRIAL: NCT05742035
Title: Quality and Biologic Characteristics of Red Blood Concentrates Obtained From Individuals With Elevated Ferritin.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Interregionale Blutspende SRK (Other)
Responsible Party: Principal Investigator, Stefano Fontana, Head of Medical Department, Principal Investigator, Interregionale Blutspende SRK
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-00274
Record Dates: First submitted 2023-02-06; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Hereditary Hemochromatosis; Hyperferritinemia
MeSH Terms: conditions — Hemochromatosis; Hyperferritinemia | interventions — Phlebotomy

STUDY DESIGN:
Intervention Model Description: Prospective inclusion of individual and group allocation according to the collected clinical data and diagnoses.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors of quality parameters don't know the diagnosis of the included participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hereditary hemochromatosis (Experimental): Individual with ferritin >500 ng/mL and documented homozygous or compound heterozygous HFE-gen mutation.
  Interventions: Procedure: Venipuncture
- secondary hyperferritinemia (Experimental): Individual with ferritin >500 ng/mL, not fulfilling the criteria for hereditary hemochromatosis.
  Interventions: Procedure: Venipuncture
- healthy blood donor with normal ferritin value. (Other): Healthy comparator.
  Interventions: Procedure: Venipuncture

INTERVENTIONS:
Procedure: Venipuncture — Bloodletting of 450 mL, followed by separation of the whole blood in 2 blood components: 1 red blood cell concentrate and 1 plasma. Measurement of the outcomes in the red blood cell concentrate.

SUMMARY:
Iron overload in hereditary hemochromatosis (HH) is treated by phlebotomy. It is unclear, if individuals with hyperferritinemia due to hereditary hemochromatosis or to secondary causes are suitable as blood donors. The study investigates hemolysis and several other quality parameters of red blood cell concentrates (RBC) obtained from 80 individual with ferritin >500 ng/mL - due to hereditary hemochromatosis or secondary - and 20 healthy blood donors as control.

DETAILED DESCRIPTION:
Iron overload in hereditary hemochromatosis is treated by phlebotomy. In Switzerland and in many other coutries, these individuals are not accepted for blood donation until ferritin values and phlebotomy intervals are in the normal range.

Individual with secondary hyperferritinemia, e. g. related to metabolic syndrome, are accepted as blood donors according to their clinical situation.

It is unclear if the quality of blood products issued from individuals with hyperferritinemia due to hereditary hemochromatosis or to secondary causes is comparable with the quality of those issued from healthy blood donors, and if their characteristics comply with the international standards.

The study investigates the hemolysis rate and several other quality parameters in RBC obtained from 80 individual with ferritin >500 ng/mL - due to hereditary hemochromatosis or secondary - and 20 healthy blood donors as control. For this purpose, whole blood donations are manufactured according to the standard processes applied in the blood bank. Several standard quality parameters as well as biologic, rheologic, and oxydative stress-related variables are measured and compared, both with the current regulations and with those of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years
* Body weight > 50 Kg
* Haemoglobin ≥ 135 g/l (males), ≥ 125 g/l (females)
* In subjects of the HH and non-HH group: ferritin values >500 ng/ml, which must have been measured in the last three months before the inclusion in the study (either at the Blood Donation service or elsewhere), not followed by a blood donation or a phlebotomy
* In subjects of the HH group: genetic test demonstrating the presence of p.C282Y homozygous or p.C282Y/p.H63D compound heterozygous HFE-gene mutation
* In subjects of the control group: ferritin values < 300 ng/ml (males) or < 200 ng/ml (females)
* Written informed consent to the participation in the study

Exclusion Criteria:

* Inadequate vein access for whole blood collection
* Body weight < 50 kg
* Chronic viral infection (hepatitis B or C, HIV)
* Previous acute coronary heart disease
* Previous or current history of epilepsy
* Other severe conditions that could significantly increase the phlebotomy risk, based on individual medical evaluation
* No informed consent
* Pregnancy (according to the information on the standard blood donor questionnaire)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Hemolysis rate vs regulatory standards. | After 42 days of storage
  To verify that the hemolysis rate in % at the end of storage (day 42) of RBC from individuals with elevated ferritin is within the current accepted European standard of 0.8%.

SECONDARY OUTCOMES:
Hemolysis hyperferritinemia vs controls end of storage. | After 42 days of storage
  Comparison of haemolysis rate in % at day 42 in RBC from individuals with elevated ferritin of any cause and those with normal ferritin levels.
Hemolysis hereditary hemochromatosis (HH) vs secondary hyperferritinemia entd of storage. | After 42 days of storage
  Comparisons of hemolysis rate in % at day 42 in RBC from individuals with HH and those with secondary hyperferritinemia.
Hemolysis hyperferritinemia vs controls day 1. | After 42 days of storage
  Comparisons of hemolysis rate in % at day 1 in RBC from individuals with hyperferritinemia and those with normal ferritin.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Blutspendedienst SRK beider Basel, Basel
  - Interregionale Blutspende SRK, Bern